CLINICAL TRIAL: NCT07182487
Title: Relationship Between Postural Sway of Trunk and Upper Extremity Functional Skills in Patients With Parkinson's Disease(pwPD)
Brief Title: Postural Sway of Trunk and Upper Extremity Functional Skills in Atient With Parkinson Disease (pwPD)
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: Gyko
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: PARKINSON DISEASE (Disorder); Postural Instability; Trunk Stability Impairment; Upper Extremity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Individuals between the ages of 40 and 75 diagnosed with idiopathic Parkinson's disease (n=40±5)
- 2: Healthy individuals between the ages of 40-75 (n=40±5)

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease, characterized clinically by motor and non-motor symptoms, including bradykinesia, resting tremor, and/or rigidity. Among the motor deficits observed in PD, decreased postural control often results in decreased balance. Furthermore, losses in many upper extremity and manual skills are also observed in PD. Loss of postural control is one of the key motor symptoms observed in the advanced stages of PD, increasing the risk of falls. Analysis of postural control deficits is critical for assessing disease progression and treatment planning in PD. In this context, gyroscope-based motion analysis systems are used as a reliable method for assessing trunk sway.Sensory deficits, such as decreased spatial and temporal tactile discrimination thresholds in the fingertips, are also observed in PD. Reaching and grasping deficits are more common when patients have significant difficulty initiating movements toward a target. These patients exhibit deficits in manipulating the hand relative to object geometry. A loss of coordination between reach and grasp timing is observed. These patients generally rely on visual cues to control movement. They experience difficulties in optimal object manipulation due to difficulties planning finger placement.Studies have shown a strong relationship between postural control and fine motor functions. For high-quality distal movement, better proximal stabilization is necessary. During upper extremity functions, the body's center of gravity must shift with arm movements, allowing adaptation to changing gravity. Good trunk control is essential for this dynamic process of maintaining balance. Studies examining this link between trunk control, balance, and hand functions are available in the literature. Among these studies conducted in diverse populations, studies involving PD are very few. In light of this information, our study was designed to investigate the relationship between postural trunk sway and hand dexterity in PD. Therefore, the aim of this study was to determine the relationship between postural sway and upper extremity functional abilities in PD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 40-75 years, diagnosed with idiopathic PD according to the UK Parkinson's Disease Association Brain Bank criteria by a specialist neurologist, with a Modified Hoehn & Yahr (m-HY) scale stage ≤4, and with a Mini Mental State Examination score of ≥22 for those with training and ≥18 for those without training, and with no known disease, volunteered to participate in the study.
* Individuals with no other known neurological and/or systemic disease
* Individuals without any upper extremity contractures

Exclusion Criteria:

* Individuals with severe balance and walking difficulties
* Individuals with diagnosed and/or treated psychiatric illnesses who are considered unable to complete the required tests
* Those taking neuroleptic medications or antidepressants
* Individuals with orthopedic conditions that interfere with manual dexterity tests, such as severe dyskinesia, carpal tunnel syndrome, tendon injuries, or finger amputations; rheumatological diseases such as rheumatoid arthritis and osteoarthritis; and individuals with any neurological disease other than PD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged between 40 and 75 years (n=40±5) who applied to the Neurology Clinic of the Faculty of Medicine of KSÜ Training and Research Hospital, diagnosed with Idiopathic Parkinson's disease (PD) by a neurologist, having stage ≤4 on the Modified Hoehn&Yahr (m-HY) scale, and having scores of ≥22 in the educated and ≥18 in the uneducated according to the Mini Mental State Examination, and healthy individuals of a similar age group (n=40±5)
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
The Gyko Device for postural truk stability | first day of the assessment
  This device, manufactured by Mikrogate and manufactured in Italy, is used as a portable inertial measurement unit for motion analysis and postural stability assessment. A sensor placed on a sling is used to analyze the displacement of the patient's center of gravity using a computer. The patient is asked to walk for 30 seconds. The data collected includes postural data such as sway length and area, sway excursion speed, and sway frequency. Studies have shown that the device has high absolute and relative reliability and provides measurements consistent with other validation methods . The device's ease of use and portability make it preferred in clinical and sports settings. Furthermore, the data accuracy it provides across different ground conditions and movement patterns has contributed to its widespread acceptance.
The 9-Hole Peg Test (DDPT) | Day 1
  The 9-Hole Peg Test (DDPT) is a validated test for PD that measures manual dexterity in seconds based on performance (21). The test material consists of nine standard-sized small rods and a nine-hole platform on which to place them. The test will be administered with the patient in a sitting position. The patient will be asked to place nine rods in the round compartment of the box as quickly as possible into the holes of the box, starting from the edge farthest from the compartment and immediately withdraw them from the edge closest to the compartment. The test will begin with the dominant hand, and the time will be measured with a stopwatch, starting when the hand touches the rods and ending when the last rod is placed in the box. The same procedure will be applied to the other hand. In this study, the arithmetic mean of the test times, repeated twice, will be recorded separately for each hand.

SECONDARY OUTCOMES:
Sosyodemographic form | Day 1
  Medical history (disease duration and symptoms), demographic information (age, height, weight, education level), habits, medications, level of dependency in mobility in daily life, use of assistive devices
Modified Hoehn & Yahr (m-HY) scale | Day 1
  PD disability will be assessed with the m-HY scale: stage 1.0 (unilateral involvement only); stage 1.5 (unilateral and axial involvement); stage 2.0 (bilateral involvement without balance impairment); stage 2.5 (mild bilateral disease with improvement in the pull test); stage 3.0 (mild to moderate bilateral disease; some postural impairment; physically independent); stage 4.0 (severe disability; still able to walk or stand unaided). Symptom severity in PD was graded using the Unified Parkinson's Disease Rating Scale (UPDRS): part I (mental dysfunction and mood); part II (activities of daily living); part III (motor component); part IV (treatment-related complications)
Unified Parkinson's Disease Rating Scale (UPDRS) | Day 1
  Symptom severity in PD is rated using the Unified Parkinson's Disease Rating Scale (UPDRS). Several items on this scale assess upper extremity and hand function. The Activities of Daily Living section assesses handwriting, cutting food, and grasping utensils. The Motor section assesses finger tapping, hand movements, and rapid alternating hand movements. These test items are scored from 0 to 4, with 4 representing maximum impairment and 0 representing normal movement ability. The UPDRS is comprised of subsections: Section I (mental dysfunction and mood); Section II (activities of daily living); Section III (motor); and Section IV (treatment-related complications).
Mini Mental State Examination(MMSE) | Day 1
  The test was developed by Folstein in 1975. Its Turkish validity and reliability study was conducted by Güngen et al. in 2002. The Mini Mental State Examination (MMSE), which assesses cognitive functions in five separate sections (orientation, registration, attention and calculation, recall, and language), is frequently used and is quite suitable for screening cognitive function in the elderly. A score below 24 on the MMSE indicates dementia, 24-26 indicates mild cognitive impairment, and 26 or above indicates normal cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Study Chair — Kahramanmaras Sutcu Imam University; Yusuf Şinasi Kırmacı, Asisstant Prof, Principal Investigator — Kahramanmaras Sutcu Imam University; Asiya Uzun, Asisstant Prof, Study Chair — Kahramanmaras Sutcu Imam University; Abdulkadir Ertürk, Msc, Study Chair — Kahramanmaras Sutcu Imam University; Tuğçe Simay Özbay, Msc, Study Chair — Kahramanmaras Sutcu Imam University; Buket Tuğan Yıldız, Associate Professor, Study Chair — Kahramanmaras Sutcu Imam University; Deniz Tuncel Berktaş, Proffessor, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)